CLINICAL TRIAL: NCT02428231
Title: A Multicenter, Treatment-Blind Phase 3b Study to Evaluate Whether 6-Week Up-Titration in Tecfidera® Dose is Effective in Reducing the Incidence of Gastrointestinal Adverse Events in Patients With Multiple Sclerosis
Brief Title: Tecfidera Slow-Titration Study
Acronym: TITRATION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS416; 2014-004562-22 (EudraCT Number)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment (One-Week Titration) (Active Comparator): 120 mg DMF twice daily for 1 week, then 240 mg (as 2 120-mg capsules) DMF twice daily for 11 weeks
  Interventions: Drug: dimethyl fumarate
- Slow Up-Titration (Six-Week Titration) (Experimental): 120 mg DMF once daily (morning dose) and placebo once daily (evening dose) for 2 weeks, then 120 mg DMF twice daily for 2 weeks, then 240 mg (as 2 120-mg capsules) DMF in the morning and 120 mg in the evening for 2 weeks, then 240 mg (as 2 120-mg capsules) DMF twice daily for 6 weeks
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Participants will be dosed twice daily for 12 weeks.
  Other Names: DMF; Tecfidera; BG00012

SUMMARY:
The primary objective of the study is to assess whether a 6-week titration (compared with a 1-week titration) is effective in reducing the incidence of dimethyl fumarate (DMF [Tecfidera])-related gastrointestinal (GI) adverse events (AEs) in participants with multiple sclerosis (MS). The secondary objective of this study is to assess whether a 6-week titration (compared with a 1-week titration) is effective in reducing the average severity and duration of GI symptoms over 12 weeks of DMF treatment in this study population.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of MS consistent with locally labeled indication for DMF
* No prior treatment with DMF
* Female subjects of childbearing potential who are not surgically sterile and male subjects must practice effective contraception during their participation in the study
* Have had a recent complete blood count (CBC), including lymphocyte count, that does not preclude participation in the study, in the judgement of the investigator

Key Exclusion Criteria:

* Have a recent history or ongoing GI illness (e.g., peptic ulcer, irritable bowel syndrome) or any other current condition with GI signs and symptoms (e.g., nausea, vomiting, abdominal pain, or diarrhea) that may interfere with assessment of study endpoints
* Have other major comorbid conditions that preclude participation in the study, as determined by the investigator
* Participant is pregnant, breastfeeding, or planning a pregnancy during the study period
* Are receiving concomitant disease-modifying therapies for MS including, but not limited to, natalizumab, interferon beta, glatiramer acetate, fingolimod, alemtuzumab, teriflunomide, or laquinimod at screening
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity
* NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (20):
- United States (15):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Long Beach, California
  - Research Site, Miami, Florida
  - Research Site, Avon, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Lewiston, Maine
  - Research Site, Asheville, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dallas, Texas
  - Research Site, Wenatchee, Washington
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Wilrijk
- Research Site, Prague, Czechia
- Italy (2):
  - Research Site, Merano, Bolzano
  - Research Site, Montichiari

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment (One-Week Titration): Following a 2-week placebo run-in baseline period, 120 mg dimethyl fumarate (DMF) twice daily for 1 week, then 240 mg (as 2 120-mg capsules) DMF twice daily for 11 weeks.
- Slow Up-Titration (Six-Week Titration): Following a 2-week placebo run-in baseline period, 120 mg DMF once daily (morning dose) and placebo once daily (evening dose) for 2 weeks, then 120 mg DMF twice daily for 2 weeks, then 240 mg (as 2 120-mg capsules) DMF in the morning and 120 mg in the evening for 2 weeks, then 240 mg (as two 120-mg capsules) DMF twice daily for 6 weeks.
Period: Overall Study
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration)
Started | 30 | 32
Completed | 17 | 15
Not Completed | 13 | 17
Not completed — Other | 10 | 16
Not completed — Required Symptomatic Therapy | 0 | 1
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Treatment (One-Week Titration): Following a 2-week placebo run-in baseline period, 120 mg DMF twice daily for 1 week, then 240 mg (as 2 120-mg capsules) DMF twice daily for 11 weeks.
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration) | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.77) | 42.5 (11.12) | 44.0 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With a Worsening in Severity of Gastrointestinal (GI) Adverse Events (AEs) on the Gastrointestinal Symptom Rating Scale (GSRS)
Description: The GSRS is a weekly recall scale to rate the severity of GI symptoms in participants. It was modified for daily recall in this study. GSRS is a rating scale consisting of 15 items for assessment of GI symptoms (see Appendix 1). Items are scored for intensity on a 7-grade Likert scale, defined by descriptive anchors such that 0 = none, 1 = minor, 2 = mild, 3 =moderate, 4 = moderately severe, 5 = severe, and 6 = very severe discomfort. The overall GSRS score is the mean of these 15 items, varying from 0 to 6; a score of 0 indicates that no symptoms are present, and a score of 6 indicates the worst possible degree of all symptoms. A higher score relative to Baseline indicates worsening of severity.
Time Frame: from Week 2 (Baseline) to Week 14
Population: The limited number of participants enrolled and the early termination of the study resulted in efficacy data not collected, and efficacy outcomes not analyzed, as per the pre-specified plan of analysis.
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Average Change From Baseline in GSRS Scores During DMF Treatment
Description: Average change from baseline in GSRS scores over the 12 weeks of DMF treatment as measured by the total change in GSRS scores from baseline divided by the total number of days with GSRS scores recorded. The GSRS is a weekly recall scale to rate the severity of GI symptoms in participants. It was modified for daily recall in this study. GSRS is a rating scale consisting of 15 items for assessment of GI symptoms (see Appendix 1). Items are scored for intensity on a 7-grade Likert scale, defined by descriptive anchors such that 0 = none, 1 = minor, 2 = mild, 3 =moderate, 4 = moderately severe, 5 = severe, and 6 = very severe discomfort. The overall GSRS score is the mean of these 15 items, varying from 0 to 6; a score of 0 indicates that no symptoms are present, and a score of 6 indicates the worst possible degree of all symptoms.
Time Frame: Week 2 (Baseline), Week 14
Population: as for outcome 1
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to First Worsening From Baseline in GSRS Score
Description: The GSRS is a weekly recall scale to rate the severity of GI symptoms in participants. The GSRS is a weekly recall scale to rate the severity of GI symptoms in participants. It was modified for daily recall in this study. GSRS is a rating scale consisting of 15 items for assessment of GI symptoms (see Appendix 1). Items are scored for intensity on a 7-grade Likert scale, defined by descriptive anchors such that 0 = none, 1 = minor, 2 = mild, 3 =moderate, 4 = moderately severe, 5 = severe, and 6 = very severe discomfort. The overall GSRS score is the mean of these 15 items, varying from 0 to 6; a score of 0 indicates that no symptoms are present, and a score of 6 indicates the worst possible degree of all symptoms. A higher score relative to Baseline indicates worsening of severity.
Time Frame: Week 2 (Baseline), Week 14
Population: as for outcome 1
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Recovery to Baseline From Last Occurrence of Worst GSRS Score
Description: as for outcome 3
Time Frame: Week 2 (Baseline), Week 14
Population: as for outcome 1
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Average Change From Baseline in GSRS Scores to the End of Weeks 4, 6, 8, 10, 12, and 14
Description: Average change from baseline to end of DMF treatment in the GSRS. The GSRS is a weekly recall scale to rate the severity of GI symptoms in participants. It was modified for daily recall in this study. GSRS is a rating scale consisting of 15 items for assessment of GI symptoms (see Appendix 1). Items are scored for intensity on a 7-grade Likert scale, defined by descriptive anchors such that 0 = none, 1 = minor, 2 = mild, 3 =moderate, 4 = moderately severe, 5 = severe, and 6 = very severe discomfort. The overall GSRS score is the mean of these 15 items, varying from 0 to 6; a score of 0 indicates that no symptoms are present, and a score of 6 indicates the worst possible degree of all symptoms.
Time Frame: Week 2 (Baseline), Weeks 4, 6, 8, 10, 12, 14
Population: as for outcome 1
Arm/Group | Standard Treatment (One-Week Titration) | Slow Up-Titration (Six-Week Titration)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study through Week 14 plus 2 weeks (±5 days) follow-up. Serious events were collected from time of informed consent and non-serious events were collected from the first dose and throughout the study.
Groups:
- Standard 1-Week Titration Arm: Following a 2-week placebo run-in baseline period, 120 mg DMF twice daily for 1 week, then 240 mg (as 2 120-mg capsules) DMF twice daily for 11 weeks.
- 6-Week Titration Arm: Following a 2-week placebo run-in baseline period, 120 mg DMF once daily (morning dose) and placebo once daily (evening dose) for 2 weeks, then 120 mg DMF twice daily for 2 weeks, then 240 mg (as 2 120-mg capsules) DMF in the morning and 120 mg in the evening for 2 weeks, then 240 mg (as two 120-mg capsules) DMF twice daily for 6 weeks.
Arm/Group | Standard 1-Week Titration Arm | 6-Week Titration Arm
Serious Adverse Events (participants affected / at risk) | 2/30 | 1/32
Other Adverse Events (participants affected / at risk) | 18/30 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard 1-Week Titration Arm (N=30) | 6-Week Titration Arm (N=32)
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard 1-Week Titration Arm (N=30) | 6-Week Titration Arm (N=32)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Cystitis (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 4
Multiple sclerosis relapse (Nervous system disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Flushing (Vascular disorders) | 7 | 6

LIMITATIONS AND CAVEATS:
The Sponsor decided to terminate the study as a result of an evaluation of ongoing development programs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.